CLINICAL TRIAL: NCT00672828
Title: Promoting Colon Cancer Screening Among African Americans
Brief Title: Interactive Computer Program or Brochure in Increasing Colorectal Cancer Screening Among African Americans
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUSN-0604-01B; CDR0000584262 (Registry Identifier: PDQ (Physician Data Query)); 5R01CA115983-05 (NIH)
Record Dates: First submitted 2008-05-03; First posted 2008-05-06 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-tailored CRC screening brochure (Active Comparator): Participants undergo a baseline interview via telephone and receive a non-tailored CRC screening brochure in the clinic prior to visit with healthcare provider. Participants then undergo telephone interviews at 1 week, 6 months, and 15 months.
  Interventions: Behavioral: Non-tailored CRC screening brochure
- Interactive computer intervention (Experimental): Participants undergo a baseline interview via telephone and complete an interactive computer intervention in the clinic prior to visit with healthcare provider. Participants then undergo telephone interviews at 1 week, 6 months, and 15 months.
  Interventions: Behavioral: Interactive computer intervention

INTERVENTIONS:
Behavioral: Non-tailored CRC screening brochure — Patients receive written educational material about colorectal cancer and prompting to talk to their doctor about getting tested.
  Arms: Non-tailored CRC screening brochure
Behavioral: Interactive computer intervention
  Arms: Interactive computer intervention

SUMMARY:
RATIONALE: An interactive computer program may be more effective than a brochure in increasing colorectal cancer screening among African Americans.

PURPOSE: This randomized clinical trial is studying an interactive computer program to see how well it works compared with a brochure in increasing colorectal cancer screening among African Americans.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare rates of participation in fecal occult blood testing and endoscopic screening (colonoscopy or sigmoidoscopy) among African-Americans who receive an interactive computer intervention (ICI) versus a non-tailored colorectal cancer screening brochure.
* Examine mediators and moderators of intervention effectiveness as depicted in the conceptual model.

OUTLINE: This is a multicenter study.

Participants are stratified according to site, age (≤ 65 years old vs > 65 years old) and gender. Participants are randomized to one of two arms.

* Arm I (non-tailored colorectal cancer screening brochure): Participants undergo a baseline interview via telephone and receive a colorectal cancer screening brochure in the clinic prior to visit with healthcare provider. Participants then undergo telephone interviews at 1 week, 6 months, and 15 months.
* Arm II (interactive computer intervention [ICI]): Participants undergo a baseline interview via telephone and complete an ICI in the clinic prior to visit with healthcare provider. Participants then undergo telephone interviews at 1 week, 6 months, and 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently being seen in the primary care clinics of Wishard Memorial Hospital (Indianapolis, IN), Roudebush Veterans Affairs Medical Center (Indianapolis, IN), IU Health Family Medicine Center (Indianapolis, IN) or Norton Louisville Primary Care Clinic (Louisville, KY)
* African-American who is currently non-adherent to screening guidelines, meeting all of the following criteria:

  * No fecal occult blood test in the past 12 months
  * No sigmoidoscopy in the past 5 years
  * No colonoscopy in the past 10 years
* Patients with average and increased risk for colorectal cancer are eligible
* No personal history of colorectal cancer

PATIENT CHARACTERISTICS:

* Participants must have a telephone
* English-speaking
* Able to read at a 5th grade reading level
* No medical condition that prohibits colorectal cancer screening

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 51 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Self-reported colorectal cancer (CRC) screening adherence with medical record verification of screening test completion | 6 and 15 months post-intervention

SECONDARY OUTCOMES:
Self-reported CRC discussion and screening test recommendation from provider on intervention/clinic visit date | 1 week post-intervention
  Discussion of Fecal Occult Blood Test (FOBT), colonoscopy, and sigmoidoscopy is assessed. Participants report on whether or not an FOBT kit was given to them during this visit. Additionally, participants report on whether or not someone in the doctor's office made an appointment for a colonoscopy or sigmoidoscopy.
Provider documentation of CRC discussion and screening test recommendation on intervention/clinic visit date | 1 week post-intervention
  Medical record documentation of discussion of FOBT, providing participant with an FOBT kit, discussion and/or ordering a colonoscopy, and discussion and/or ordering a sigmoidoscopy is assessed.
Self-reported CRC health beliefs | Pre-intervention (baseline),1 week post-intervention, and 6 months post-intervention
  Changes in perceived risk, benefits to screening, barriers to screening, and self-efficacy for CRC screening are assessed.
Self-reported stage of CRC screening test adoption | Pre-intervention (baseline),1 week post-intervention, 6 months post-intervention, and 15 months post-intervention
  For FOBT, colonoscopy, and sigmoidoscopy, stage of adoption measured as either precontemplation, contemplation, preparation, action, or maintenance.

OTHER OUTCOMES:
Patient characteristics as CRC screening predictors | Pre-intervention (baseline), intervention date, 1 week post-intervention, 6 months post-intervention, and/or 15 months post-intervention
  Age, gender, marital status, education, health literacy, income, employment, insurance coverage, BMI, co-morbidities, family history of cancer, family or friend encouragement to have CRC screening, CRC knowledge, physician trust, fatalism views, and health temporal orientation are assessed.
Clinic variables as CRC screening predictors | Pre-intervention (baseline), 1 week post-intervention, 6 months post-intervention, and 15 months post-intervention
  Clinic site, participant's reason for health care provider visit, and prior recommendation(s) to do CRC screening are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rawl, PhD, RN, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Rawl SM, Christy SM, Perkins SM, Tong Y, Krier C, Wang HL, Huang AM, Laury E, Rhyant B, Lloyd F, Willis DR, Imperiale TF, Myers LJ, Springston J, Skinner CS, Champion VL. Computer-tailored intervention increases colorectal cancer screening among low-income African Americans in primary care: Results of a randomized trial. Prev Med. 2021 Apr;145:106449. doi: 10.1016/j.ypmed.2021.106449. Epub 2021 Feb 4. PMID 33549682
- [Derived] Christy SM, Perkins SM, Tong Y, Krier C, Champion VL, Skinner CS, Springston JK, Imperiale TF, Rawl SM. Promoting colorectal cancer screening discussion: a randomized controlled trial. Am J Prev Med. 2013 Apr;44(4):325-329. doi: 10.1016/j.amepre.2012.11.032. PMID 23498096